CLINICAL TRIAL: NCT05321147
Title: A Multi-center Phase Ib Trial Evaluating the Safety and Efficacy of Lacutamab in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma That Express KIR3DL2
Brief Title: Safety and Efficacy of Lacutamab in Patients With Relapsed/Refractory Peripheral T-cell Lymphoma That Express KIR3DL2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH4102-102
Record Dates: First submitted 2022-04-04; First posted 2022-04-11 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Peripheral T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTCL that express KIR3DL2 (Experimental): lacutamab will be administered every week for 5 weeks then every 2 weeks for 10 administrations then every 4 weeks until disease progression or unacceptable toxicity.
  Interventions: Biological: lacutamab

INTERVENTIONS:
Biological: lacutamab — Patients will receive a fixed dose of 750mg as 1-hour IV infusion
  Other Names: IPH4102

SUMMARY:
This is a multi-center phase Ib study, which evaluates the safety and efficacy of lacutamab monotherapy in patients with relapsed/refractory peripheral T-cell lymphoma that express KIR3DL2.

DETAILED DESCRIPTION:
This is an open-label, single-arm multicenter study. Eligible patients will be enrolled and will receive fixed dose of 750mg Lacutamab as a 1-hour IV infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Any subtype of PTCL;
2. Patients should have received at least one prior line of systemic therapy;
3. Patient with documented refractory, relapsed, or progressive disease. Patients must receive at least 2 cycles of prior line of systemic therapy (N-1). The patients who have withdrawn from prior (N-1) line of systemic therapy due to unacceptable toxicity must have received at least 2 cycles of prior (N-2) line of therapy;
4. KIR3DL2 expression (≥ 1%) based on central evaluation by IHC of either a newly acquired biopsy (preferred) or a tissue sample collected from a historical lymph node biopsy;
5. Presence of at least 1 target lesion on PET/CT scan at screening;
6. Male or Female, at least 18 years of age;
7. ECOG performance status ≤ 2;
8. The patient must have a minimum wash-out period of 3 weeks between the last dose of prior line of systemic therapy and first dose of lacutamab;
9. Patients should have recovered from clinically relevant adverse events related to prior therapy to ≤ grade 1. Certain toxicities will not be considered in this category (e.g., Grade 2 alopecia, peripheral neuropathy and/or endocrine end-organ failure being adequately managed by hormone replacement therapy);
10. Adequate baseline laboratory data:

    Hematology:
    * Hemoglobin >9 g/dL
    * Absolute neutrophil count (ANC) ≥1,000/µL,
    * Platelets ≥50,000/µL,

    Biochemistry:
    * Bilirubin ≤1.5 X upper limit of normal (ULN) or ≤3 X ULN for patients with Gilbert's disease,
    * Serum creatinine ≤1.5 X ULN,
    * Creatinine clearance ≥30 mL/min, assessed using the Cockcroft & Gault formula
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤3 X ULN;
11. Women of childbearing potential (WOCBP): Premenopausal females who had at least one menstrual cycle in the past 12 months and capable to become pregnant. They must have a negative serum beta-HCG pregnancy test result within seven days before start of treatment;
12. Women of childbearing potential and all men (and their female partners of childbearing potential) who are sexually active must agree to use adequate method of contraception at study entry, during treatment and for at least 9 months (270 days) following the last dose of study drug
13. Signed informed consent form prior to any protocol-specific procedure being performed.

Exclusion Criteria:

1. Treatment with > 8 lines of systemic therapies prior to enrollment. Consolidation therapy including stem cell transplant is not considered a line of therapy;
2. Patients having a life expectancy of less than 3 months;
3. Receipt of live vaccines within 4 weeks prior to treatment;
4. Known central nervous system (CNS) lymphoma involvement;
5. Prior treatment with lacutamab;
6. Concurrent enrollment in another clinical trial, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study;
7. Concomitant administration of radiotherapy or systemic anti-cancer therapy including but not restricted to: chemotherapy, biological agents or immunotherapy;
8. Autologous stem cell transplantation less than 3 months prior to enrollment;
9. Prior allogenic transplantation;
10. Patients who have undergone major surgery ≤ 4 weeks prior to study entry;
11. Patients with known NCI-CTCAE grade 3 or higher active systemic or cutaneous viral, bacterial, or fungal infection;
12. Patients who have active Hepatitis B or C virus infection confirmed by PCR;
13. Patients known or tested positive for human immunodeficiency virus (HIV);
14. Patients with a history of other malignancies during the past three years apart from the disease subject of this study. The following are exempt from the three-year limit: non_melanoma skin cancer, lymphomatoid papulosis, resected thyroid cancer, biopsy-proven cervical intraepithelial neoplasia, Ductal carcinoma in situ (DCIS) or cervical carcinoma in situ.
15. Pregnant or breastfeeding women;
16. Patients with congestive heart failure, Class III or IV, by New York Heart Association (NYHA) criteria;
17. Patients with any serious underlying medical condition that would impair their ability to receive or tolerate the planned treatment and/or comply with study protocol;
18. Patients with dementia or altered mental status that would preclude understanding and rendering of informed consent document.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs) | From consent is obtained until EOT visit (28 days after the last administration of study drug lacutamab)
  Frequency and intensity of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (10):
  - University of Alabama at Birmingham- O'Neal Comprehensive Cancer Center, Birmingham, Alabama
  - University of California at Irvine - Chao Family Comprehensive Cancer Center, Orange, California
  - Goshen Health- Goshen Hospital, Goshen, Indiana
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center- David H. Koch Center for Cancer Care, New York, New York
  - Allegheny Health, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Health Hollings Cancer Center, Charleston, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- South Korea (10):
  - Inje University Busan Paik Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul